CLINICAL TRIAL: NCT02114775
Title: Growth Hormone or Sildenafil as Therapies for Fatigue in MTBI
Brief Title: Growth Hormone or Sildenafil as Therapies for Fatigue in Mild- Traumatic-brain-injury (MTBI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 13-0324
Record Dates: First submitted 2014-01-31; First posted 2014-04-15 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Traumatic Brain Injury
Keywords: mild traumatic brain injury; growth hormone; fatigue; sildenafil; neurology
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Fatigue | interventions — Growth Hormone; Human Growth Hormone; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recombinant Growth Hormone (Active Comparator): Double blind placebo/Genotropin cross over design for 6 months with cross over at 3 months. Then open label Genotropin from month 6 - 12.
  Interventions: Drug: Growth Hormone; Drug: Placebo
- Sildenafil (Active Comparator): Double blinded placebo/Sildenafil crossover design for 6 months with crossover at month 3. Then open label Sildenafil from months 6-12.
  Interventions: Drug: Sildenafil; Drug: Placebo

INTERVENTIONS:
Drug: Growth Hormone — 0.4 mg/day injected subcutaneously for one month then increased to 0.6 mg/day for two months during crossover phase. After crossover phase, 0.6 mg/day for six months
  Other Names: Genotropin
  Arms: Recombinant Growth Hormone
Drug: Sildenafil — 50 mg by mouth daily
  Other Names: Viagra
  Arms: Sildenafil
Drug: Placebo — Placebo either injected (GH group) or orally (sildenafil group) daily for three months during crossover phase of the study

SUMMARY:
The overall goal is to determine whether perceptual or performance fatigue can be reduced in MTBI patients with and without growth hormone (GH) deficiency by treating them in a crossover fashion based upon GH status.

A battery of functional, fatigue, cognitive, imaging and blood flow tests will be performed to assess the efficacy of the two drug interventions, Growth hormone and Sildenafil.

DETAILED DESCRIPTION:
Three primary outcome measures are proposed:

1. Perceptual fatigue as measured weekly using the Brief Fatigue Inventory (BFI) (59).
2. Performance fatigue as measured at baseline and month 3, 6 and 12 using hand and leg dynamometry.
3. Neuropsychological function as measured at baseline and month 12.

Secondary outcomes will include:

1. Modified 6 minute walk performance as measured at baseline, and month 3, 6 and 12.
2. Mood and quality of life using the Profile of Mood States, Quality of Life Assessment of GH Deficiency in Adults questionnaire, and a grief assessment (60) (POMS), measured at baseline, and month 3, 6, and 12.
3. Sleep quality using the Pittsburgh Sleep Quality Index (PSQI), baseline, and month 3, 6, and 12.
4. Multidimensional fatigue using Multidimensional Fatigue Symptom Inventory (MFSI) at baseline, and month 3, 6 and 12.
5. Skeletal muscle mass, as derived from lean body mass determinations, using dual energy X-ray absorptiometry (iDEXA) at baseline, and month 3, 6, and 12.
6. Physical Activity, measured daily using accelerometry.
7. Cerebral blood oxygen saturation measured at baseline and month 12.
8. Leg blood flow measured at baseline, and month 3, 6 and 12.
9. Blood Hormones at baseline and month 3, 6 and 12.
10. Characterization of brain tissue using structural, "resting state" and diffusion functional MR at baseline and month 3, 6, and 12.
11. Indirect calorimetry measured at baseline and month 3, 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

Male or female with a diagnosis of mild TBI and 6 month post-injury. Age 18 to 60 years. Complaint of fatigue, with score of 3 or greater on questions 1, 2, or 3 of the Brief Fatigue Inventory.

Exclusion Criteria:

Exclusion criteria (general)

1. Significant heart, liver, kidney, blood or respiratory disease.
2. Active coronary disease.
3. Pregnancy.
4. Alcohol or drug abuse.
5. Unable to walk unassisted.
6. Diabetes mellitus and anterior pituitary abnormalities diagnosed upon screening.
7. Premorbid history of psychiatric disorder.
8. Premorbid history of head trauma.

Exclusion criteria (sildenafil/placebo group)

1. Use of nitrates.
2. Use of alpha blockers.
3. Systolic blood pressure <100 or >150, diastolic blood pressure <60 or >90. This range is smaller than the acceptable range stated in the prescribing information for sildenafil (>90/50 and <170/110).
4. Peripheral vascular disease.
5. Use of a phosphodiesterase 5 inhibitor.

Exclusion criteria (growth hormone/placebo group)

1. Coumadin because of the risk of bleeding with daily injections of Recombinant Human Growth Hormone (rhGH) in the growth hormone (GH) arm of the study.
2. Subjects who are deficient in cortisol or thyroid at screening will be excluded until hormone abnormalities have been corrected.
3. Subjects with chronic pain who are being managed with narcotics will be excluded as the effects of central nervous system depressants may interfere with study test results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Performance fatigue as measured by using hand grip dynamometry at baseline | baseline
  Hand grip exercises will be used to measure performance fatigue at baseline
Performance fatigue as measured by using hand grip dynamometry at 3 months | 3 months
  Hand grip exercises will be used to measure performance fatigue after 3 months of study intervention
Performance fatigue as measured by using hand grip dynamometry at 6 months | 6 months
  Hand grip exercises will be used to measure performance fatigue after 6 months of study intervention
Performance fatigue as measured by using hand grip dynamometry at 12 months | 12 months
  Hand grip exercises will be used to measure performance fatigue after 12 months of study intervention
Performance fatigue as measured by using leg dynamometry at baseline | baseline
  Leg exercises will be used to measure performance fatigue at baseline
Performance fatigue as measured by using leg dynamometry at 3 months | 3 months
  Leg exercises will be used to measure performance fatigue after 3 months of study intervention.
Performance fatigue as measured by using leg dynamometry at 6 months | 6 months
  Leg exercises will be used to measure performance fatigue after 6 months of study intervention.
Performance fatigue as measured by using leg dynamometry at 12 months | 12 months
  Leg exercises will be used to measure performance fatigue after 12 months of study

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Urban, MD, Principal Investigator — University of Texas; Melinda Sheffield-Moore, PhD, Principal Investigator — University of Texas; Brent Masel, MD, Principal Investigator — Transitional Learning Center
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States